CLINICAL TRIAL: NCT04371601
Title: Safety and Effectiveness of Mesenchymal Stem Cells in the Treatment of Pneumonia of Coronavirus Disease 2019
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fuzhou General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSC-CoViD-2020
Record Dates: First submitted 2020-03-25; First posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-03

CONDITIONS: COVID-19 Pneumonia
MeSH Terms: interventions — Oseltamivir; Hormones; Oxygen Inhalation Therapy

STUDY DESIGN:
Intervention Model Description: Control group: conventional symptomatic treatments such as antiviral (oseltamivir), hormones, oxygen therapy, mechanical ventilation and other supportive therapies; Experimental group: On the basis of the above-mentioned conventional symptomatic treatment and supportive therapy, umbilical cord mesenchymal stem cells were given at 106 / Kg body weight / time, once every 4 days for a total of 4 times. Peripheral intravenous infusion was given within 3 days of first admission.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): conventional symptomatic treatments such as antiviral (oseltamivir), hormones, oxygen therapy, mechanical ventilation and other supportive therapies
  Interventions: Drug: Oseltamivir; Drug: hormones; Device: oxygen therapy
- Experimental group (Experimental): On the basis of the above-mentioned conventional symptomatic treatment and supportive therapy, umbilical cord mesenchymal stem cells were given at 106/Kg body weight / time, once every 4 days for a total of 4 times. Peripheral intravenous infusion was given within 3 days of first admission
  Interventions: Drug: Oseltamivir; Drug: hormones; Device: oxygen therapy; Procedure: mesenchymal stem cells

INTERVENTIONS:
Drug: Oseltamivir — Oseltamivir capsules
Drug: hormones — a moderate amount of hormone
Device: oxygen therapy — oxygen therapy,mechanical ventilation and other supportive therapies
Procedure: mesenchymal stem cells — mesenchymal stem cells
  Arms: Experimental group

SUMMARY:
The outbreak of coronavirus disease 2019 (COVID-19) at the end of 2019 has seen numerous patients experiencing severe acute lung injury (ALI), which developed into severe respiratory distress syndrome (ARDS). The mortality was as high as 20% -40%. Due to the lack of effective antiviral treatments, supporting treatment is the predominant therapy for COVID-19 pneumonia. Its cure is essentially dependent on the patient's immunity. While the immune system eliminates the virus, numerous inflammatory cytokines are produced and a cytokine storm occurs in severe cases.

Mesenchymal stem cells (MSCs) play an important role in injury repair and immune regulation, showing advantageous prospects in the treatment of COVID-19 pneumonia. MSCs prevent cytokine storms by retarding the TNF-α pathway, alleviate sepsis by modulating macrophages, neutrophils, NK cells, DC cells, T lymphocytes and B lymphocytes. After infused, MSCs aggregate in the lungs, improve the lung microenvironment, protect alveolar epithelia, and improve pulmonary fibrosis and pulmonary function.

DETAILED DESCRIPTION:
In vitro, Mesenchymal stem cells were revealed to inhibit the secretion of inflammatory cytokines by spleen lymphocytes and up-regulate regulatory T cells, thereby inhibiting the secretion of interferon-γ(IFN-γ) induced by lymphocytes and Tumor Necrosis Factor(TNF) induced by macrophage.

Animal models and preclinical studies have shown that mesenchymal stem cells (MSCs) were implanted into inflammatory lung tissues after infusion, which significantly improved the clinical manifestations and histopathological lesions caused by acute lung injury. Mesenchymal stem cells inhibited the effects of interleukin-1 (IL-1) through regulatory T cells (CD4 + CD25 + FOXP3 + Treg cells) and by antagonizing the expression interleukin-1 receptor (IL1-RA). Mesenchymal stem cells significantly down-regulated pro-inflammatory factors by inhibiting the expression of IL-1, TNF and IFN-γ in lung tissue, and up-regulated anti-inflammatory factor by enhancing the expression of IL -10 and regulatory T cells, respectively, thereby dampening the inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

* patients with severe COVID-19 pneumonia
* willing to give informed consent

Exclusion Criteria:

* patients with mild COVID-19 pneumonia
* liver dysfunction
* concomitant with other active infection
* renal dysfunction
* Heart failure >grade 2
* pregnant
* history of COPD

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of oxygenation index (PaO2/FiO2) ,blood gas test | 12 months
  Improvement of pulmonary function

SECONDARY OUTCOMES:
Detection of TNF-α levels, IL-10 levels | 1,3,6,12months
  Cytokines level
Detection of immune cells that secret cytokines, including CXCR3+, CD4+, CD8+, NK+ cells, and regulatory T cells (CD4 + CD25 + FOXP3 + Treg cells). | 1,3,6,12months
  Immunological status
Changes of oxygenation index (PaO2/FiO2) ,blood gas test | 1,3,6months
  Improvement of pulmonary function
Changes of c-reactive protein and calcitonin | 1,3,6,12months
  Infection biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Jianming Tan Tan, M.D and Ph.D, Study Chair — Fuzhou General Hospital
Locations (1):
- Fuzhou General Hospital, Fuzhou, Fujian, China